CLINICAL TRIAL: NCT04552795
Title: Pilot Study to Investigate the Safety and Feasibility of AntiRetroviral Therapy for Alzheimer's Disease (ART-AD)
Brief Title: Pilot Study to Investigate the Safety and Feasibility of AntiRetroviral Therapy for Alzheimer's Disease
Acronym: ART-AD
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: The University of Texas Health Science Center at San Antonio (Other)
Collaborators: Owens Medical Research Foundation (Other)
Responsible Party: Principal Investigator, Bess Frost, PhD, Associate Professor, Sam and Ann Barshop Instititute for Aging and Longevity Studies, Glenn Biggs Institute for Alzheimer's and Neurodegenerative Disorders, Department of Cell Systems and Anatomy, The University of Texas Health Science Center at San Antonio
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: HSC20200396H
Record Dates: First submitted 2020-08-11; First posted 2020-09-17 (Actual); Results first posted 2024-08-09 (Actual); Last update posted 2024-08-09 (Actual); Status verified 2024-07

CONDITIONS: Alzheimer Disease, Early Onset
MeSH Terms: conditions — Alzheimer Disease | interventions — Lamivudine

STUDY DESIGN:
Intervention Model Description: Open-label, one arm study.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (1):
- Open-Label 3TC (Experimental): 12 subjects will receive 3TC, 300-mg, daily for 24 weeks.
  Interventions: Drug: 3TC

INTERVENTIONS:
Drug: 3TC — 12 subjects will be administered 3TC, 300mg once daily, via an oral tablet for 24 weeks.
  Other Names: Epivir; lamivudine

SUMMARY:
The objective of the study is to evaluate the ability of (-)-L-2',3'-dideoxy-3'-thiacytidine (3TC) to engage its intended target, penetrate the central nervous system (CNS), suppress neurodegeneration, and assess safety and tolerability in patients with early stage Alzheimer's disease. This study will provide the initial data on target engagement and Alzheimer's disease-relevant outcomes for future trials.

DETAILED DESCRIPTION:
This open label study of 3TC will collect initial proof-of-concept data on 3TC target engagement, CNS penetration, efficacy and safety in older adults with early stage Alzheimer's disease. If successful, data will be used to design a larger phase 2 clinical trial. The investigators aim to I) Quantify 3TC target engagement and CNS penetration, II) Determine if 3TC suppresses Alzheimer's disease-relevant outcomes, and III) Assess the safety and tolerability of 3TC in older individuals with early Alzheimer's disease. The study will consist of a screening/baseline period of 30 days pre-treatment, a 24-week open label treatment period, and a follow up visit one month following treatment. Visits to the clinic include a pre-treatment screening visit that includes a comprehensive neuropsychological exam, a tablet-based neuropsychological exam, and a blood draw. For eligible participants, a lumbar puncture will be performed on day one of treatment. Participants will visit the clinic on day one of treatment and at weeks 8, 16, and 24 of treatment to complete medication checks, physical examinations, tablet-based cognitive screening, and blood draw. At week 24 of treatment, patients will undergo a post-treatment comprehensive neuropsychological exam, a lumbar puncture to collect cerebrospinal fluid, and a blood draw. One month after the final dose of medication, participants will return to the clinic for a final safety assessment and disenrollment.

ELIGIBILITY:
Inclusion Criteria:

1. Aged 50-99 years
2. Clinical diagnosis of early Alzheimer's disease (Clinical Dementia Rating (CDR) = 0.5, Mini-Mental State Exam (MMSE) = 24-30)
3. If using drugs to treat symptoms related to Alzheimer's disease, doses must be stable for at least eight weeks prior to screening visit 1
4. Labs: Adequate blood cell counts (white blood cells: 4,000-111,000 cells per microliter (cells/mcL); absolute neutrophil count: 1,800-8,700 cells/mcL; platelets: 120-500 K/µL; hemoglobin 12.0-17.5 grams/dL); LFT's within 2x normal value; creatinine clearance test (CrCl) ≥ 50 mL/min; cholesterol (≤260 mg/dl), triglycerides≤ 400 mg/dl), and glucose control (HbA1c ≤ 8%). Prothrombin time/partial thromboplastin time/international normalized ratio (PT/PTT/INR) within normal limits
5. Body mass index (BMI) within range of 19 - 35 kg/m2
6. Must have a reliable informant or caregiver
7. Participants must have no plans to travel that interfere with study visits

Exclusion Criteria:

1. Any medical or neurologic condition (other than Alzheimer's Disease) that might be a contributing cause of the subject's cognitive impairment
2. Clinically significant unstable psychiatric illness in the past six months
3. Significant hearing, vision, or motor deficits that interfere with participation
4. Alcohol or drug abuse/dependence in the past six months
5. Stroke, transient ischemic attack, or unexplained loss of consciousness in the past six months
6. Unstable angina, myocardial infarction, advanced chronic heart failure, or clinically significant conduction abnormalities within the past six months
7. Relevant brain hemorrhage, bleeding disorder and cerebrovascular abnormalities
8. Diagnosis of HIV infection or AIDS (CD4 count < 200), HIV/Hepatitis B Virus (HBV) co-infection, HBV or human T-cell leukemia virus infection
9. History of impaired renal or liver function
10. Current use of memantine or sorbitol-containing products
11. Individuals with HIV, HBV, or who have current/previous use of Nucleoside Reverse Transcriptase Inhibitors (NRTIs) or non-NRTIs.
12. Poorly controlled blood pressure (BP) (systolic BP > 160, diastolic BP > 90 mmHg)
13. Uncontrolled diabetes (HbA1c > 8%, or the current use of insulin)
14. Significant systematic illness or infection in the past 30 days
15. Pregnant women

Ages: 50 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 12 (Actual)
Dates: Start 2021-02-15 (Actual); Primary Completion 2023-05-04 (Actual); Study Completion 2023-11-04 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Bess Frost, PhD, Principal Investigator — Univ of Texas Health Science Center at San Antonio
Locations (3):
- United States (3):
  - Glenn Biggs Institute for Alzheimer's & Neurodegenerative Diseases, San Antonio, Texas
  - Sam and Ann Barshop Institute for Longevity & Aging Studies, San Antonio, Texas
  - University of Texas Health Science Center at San Antonio, San Antonio, Texas

IPD SHARING:
Plan to Share IPD: Yes
Protocol, Published Data
Supporting Information: Study Protocol
Time Frame: After study completion, upon publication of data and on ClinicalTrials.gov 1 year after primary completion date of study.
Access Criteria: Data will be analyzed by the study investigators.

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants were recruited from University of Texas Health San Antonio outpatient clinics and through local flier/newspaper advertisements.
Groups:
- Open-Label 3TC: 12 subjects will be administered a 300mg once daily oral tablet of 3TC for 24 weeks.
Period: Overall Study
Arm/Group | Open-Label 3TC
Started | 12
Completed | 12
Not Completed | 0

BASELINE CHARACTERISTICS:
Arm/Group | Open-Label 3TC
Number analyzed (Participants) | 12
Age, Customized [Mean (Full Range); unit: years]
  Average age (min, max) | 69.4 [52 to 83]
Age, Customized [Count of Participants; unit: Participants]
  Age group: <= 65 years of age | 3
  Age group: 65 - 74 years of age | 5
  Age group: 75 - 84 years of age | 4
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 9
  Male | 3
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Race: White, non-Hispanic | 9
  Race: White, Hispanic | 1
  Race: African American | 1
  Race: Asian | 1
Education Level [Mean (Standard Deviation); unit: years] | 15.3 (2.4)
Past Medical History [Count of Participants; unit: Participants]
  <= 1 Comorbidities | 2
  2+ Comorbidities | 10
Duration of Symptoms Prior to Trial [Count of Participants; unit: Participants]
  <= 1 year | 1
  1-2 years | 2
  3+ years | 2
  Unknown | 7
Average BMI [Mean (Standard Deviation); unit: kg/m^2] | 25.2 (4.6)
Concurrent Treatment with Donepezil [Count of Participants; unit: Participants] | 7

OUTCOME MEASURES:

1. Primary Outcome: Change in Reverse Transcriptase Activity From Baseline to 24 Weeks in Plasma of Study Participants
Description: The extent of 3TC target engagement was measured by calculating the change in reverse transcriptase activity in plasma of participants at baseline compared to week 24 using a modified version of the EnzCheck Reverse Transcriptase (RT) Assay.
Time Frame: Baseline to 24 weeks
Measure: Mean (Standard Error); unit: Enzyme units
Groups:
- Open-Label 3TC: 12 subjects administered once daily 300 mg 3TC for 24 weeks
Arm/Group | Open-Label 3TC
Number analyzed (Participants) | 12
Enzyme units | -0.0074 (0.03)

2. Primary Outcome: 3TC CNS Penetration
Description: CNS penetration was calculated based on the ratio of CSF to plasma levels of 3TC after 24 weeks of 3TC using High Performance Liquid Chromatography with tandem Mass Spectrometry (HPLC/MS/MS).
Time Frame: 24 weeks
Population: Three subjects removed due to missed blood or CSF draw; one subject removed based on the ROUT method of outlier analysis.
Measure: Mean (Inter-Quartile Range); unit: ng/mL
Arm/Group | Open-Label 3TC
Number analyzed (Participants) | 7
ng/mL | 0.502 [0.0215 to 0.850]

3. Secondary Outcome: Change in Dementia Severity From Baseline to Week 24 of Treatment Based on the PACC-5 Z-score
Description: The Preclinical Alzheimer Cognitive Composite (PACC-5) score is calculated as a mean normative Z-score across five measures, including MMSE (0-30), Logical Memory Delayed Recall (0-25), Digit-Symbol Coding Test (0-93), Category Fluency, and Free and Cued Selective Reminding Test (0-96). Although typically relegated to individuals with prodromal and asymptomatic disease, the PACC-5 was included given its sensitivity to Alzheimer's disease-specific cognitive change.To calculate the Z score for each patient; the formula is Z = (x - M)/SD, where x is the patient's verbal memory raw score and M and SD are the estimates from the previous step. Positive Z values indicate scores that are greater than the mean of the pooled sample, and negative values indicate scores that are less than the pooled mean.A Z-score of zero represents the mean for this study population. Negative values mean a worse outcome than the standard population.
Time Frame: Baseline to 24 weeks
Measure: Median (Inter-Quartile Range); unit: Z-score
Groups:
- Baseline: Values prior to 3TC administration
- POST-Treatment: Values after 24 weeks of 3TC administration
Arm/Group | Baseline | POST-Treatment
Number analyzed (Participants) | 12 | 12
Z-score | -1.59 [-2 to -0.59] | -1.59 [-2 to -1.2]

4. Secondary Outcome: Incidence of Treatment-Emergent Adverse Events
Description: Incidence of adverse and serious adverse events potentially due to study drug
Time Frame: Baseline to Week 24
Measure: Count of Participants; unit: Participants
Groups:
- Open-Label 3TC: 12 subjects administered 300 mg once daily 3TC for 24 weeks.
Arm/Group | Open-Label 3TC
Number analyzed (Participants) | 12
Participants
  Gastrointestinal bleeding due to peptic ulcer | 1
  No adverse events | 11

5. Secondary Outcome: Incidence of Treatment-Emergent Abnormal Vital Signs
Description: Blood pressure, heart rate, temperature, and respiration, are measured and any significant change of any of these vital signs that show a significant change from the baseline value are reported as an event.
Time Frame: Baseline to Week 24
Measure: Number; unit: Events
Arm/Group | Open-Label 3TC
Number analyzed (Participants) | 12
Events | 0

ADVERSE EVENTS:
Time Frame: 28 weeks
Arm/Group | Open-Label 3TC
All-Cause Mortality (participants affected / at risk) | 0/12
Serious Adverse Events (participants affected / at risk) | 1/12
Other Adverse Events (participants affected / at risk) | 2/12
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Open-Label 3TC (N=12)
Gastrointestinal bleeding (Gastrointestinal disorders) | 1 (12) — Gastrointestinal bleeding due to a peptic ulcer; subject was on daily aspirin
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Open-Label 3TC (N=12)
SARS-CoV-2 Infection (Infections and infestations) | 2 (2)
Mild headache (Nervous system disorders) | 2 (2)
Mild fatigue (Nervous system disorders) | 1 (1)
Mild muscle pain (Musculoskeletal and connective tissue disorders) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2021-11-08): https://cdn.clinicaltrials.gov/large-docs/95/NCT04552795/Prot_SAP_000.pdf